CLINICAL TRIAL: NCT05337852
Title: The Effect of Emotional Freedom Technique Applied in Early Pregnancy on Nausea, Vomiting and Anxiety
Brief Title: Emotional Freedom Technique in Early Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Sinem GUVEN Santur, Graduate Student, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Inonu Universty
Record Dates: First submitted 2022-03-09; First posted 2022-04-20 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Nausea Gravidarum; Anxiety; Emotion Regulation; Vomiting of Pregnancy
Keywords: Nausea; Vomiting; Anxiety; Emotional Freedom Technique; Pregnancy
MeSH Terms: conditions — Anxiety Disorders; Emotional Regulation; Nausea; Vomiting

STUDY DESIGN:
Intervention Model Description: The randomized experiment was designed as a control study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): To the pregnant women in the experimental group;
  * Emotional freedom technique was applied online with the researcher twice a week.
  * PUQE, PRAQ-2 tests will be applied before the intervention,
  * SUE and PUQE will be applied before and after each session,
  * After 2 sessions, post-test data will be obtained with PUQE, SUE, PRAQ-2.
  Interventions: Other: Emotional Freedom Technique
- Control group (No Intervention): * After each intervention applied to the experimental group, SUE and PUQE will be applied to the control group over the phone, simultaneously.
  * After 1 week, post-test data will be obtained with PUQE, SUE, PRAQ-2.

INTERVENTIONS:
Other: Emotional Freedom Technique — To the pregnant women in the experimental group; Emotional freedom technique was applied online with the researcher twice a week. The "release protocol of EFT" was taught to the participants and it was applied between the interviews made by the researcher. Whether the participant did the application or not was confirmed by phone and a homework schedule was used for smooth follow-up.
  * PUQE, PRAQ-2 tests will be applied before the intervention,
  * SUE and PUQE will be applied before and after each session,
  * After 2 sessions, post-test data will be obtained with PUQE, SUE, PRAQ-2.
  Arms: Experimental group

SUMMARY:
One of the most common discomforts in early pregnancy is nausea and vomiting. Although its etiology is not known exactly, it affects an average of 50-90% of pregnant women. The severity of nausea-vomiting can vary from person to person, as well as in different pregnancies of the woman. The severity of nausea-vomiting is affected by hormonal, psychological and social factors. Adaptation to pregnancy, spouse relations, future anxiety and social support perception in nausea and vomiting experienced during early pregnancy affect women negatively and cause anxiety. The severity of nausea and vomiting also increases due to anxiety. As the severity of nausea-vomiting increases, the search for solutions to this situation and their applications to health institutions increase. Many non-pharmacological methods (respiratory exercises, acupuncture, acupressure, etc.) are used in treatment, as well as hydration, rest and pharmacological agents. One of these methods is the emotional liberation technique, which is included in cognitive behavioral therapies. This method basically treats the person physiologically and psychologically as a whole, similar to other cognitive behavioral therapies, unless there is a physiological disorder. It is aimed to reach a solution by raising awareness for the emotion felt, avoiding negative emotions and focusing on affirmations to replace them. Emotional liberation technique is an easy-to-apply and fast-solving technique in cases recorded in the subconscious with negative emotions and in the treatment of stress disorders in general. No use of emotional liberation technique has been found in the literature for the severity of nausea-vomiting and anxiety experienced during early pregnancy. Therefore, it is thought that this study will contribute to the literature. In addition, it is thought that this method will enrich midwifery interventions as a non-pharmacological method applied to pregnant women in the treatment of nausea-vomiting and anxiety, because this method is fast and practical, and the result is easy to reach.

The aim of this study is to determine the effect of emotional liberation technique applied during early pregnancy on nausea and vomiting severity and anxiety.

DETAILED DESCRIPTION:
Pregnancy is a process that causes physiological, psychological and social changes in the female body. Pregnancy period consists of three different trimesters, divided into three-month periods. In each trimester, different physiological and psychological processes specific to pregnancy are experienced, and different approaches specific to these processes are required for the general well-being of the woman and the healthy progression of the pregnancy.

Nausea-vomiting is one of the most common problems that occur during early pregnancy. Although its etiology is not known exactly, 50-90% of pregnant women are affected by this problem. It is thought that pregnancy hormones, gastrointestinal system disorders, hyperthyroidism, nutritional disorders and psychological factors cause nausea and vomiting or increase nausea-vomiting during early pregnancy. Nausea-vomiting in pregnancy; It is also called morning sickness, emesis gravidarum, pregnancy sickness. Nausea-vomiting during pregnancy starts on average in the 5th week of pregnancy, 8-12th week. It reaches its highest levels in the 16th weeks and is expected to decrease and disappear from the 16th week. It has been stated that the severity of nausea-vomiting during pregnancy varies from person to person, differs in each pregnancy of the person, and continues throughout the day, although it is often at the beginning of the day. Although many studies in this field focus on factors such as physiological, psychological, social and genetic, the common belief is that nausea and vomiting are based on psychological factors.

Early pregnancy symptoms such as nausea and changes in the breasts pave the way for emotional changes. In emotional changes, women generally do not feel joy for the baby during this period, but they often experience opposite feelings by wanting their pregnancy to be known by everyone. Stress and emotional changes arising from these contrasts create anxiety processes. Anxiety is defined as a disorder characterized by fear, restlessness, restlessness, tension, and changes such as sweating, dyspnea, and sleep problems experienced for an unknown or unidentified reason. Anxiety disorders are more common in women than men, and anxiety disorders can be seen in 30% of women in their reproductive years. Studies have shown that the rate of anxiety disorders during pregnancy varies between 6% and 30%. Among the causes of anxiety in pregnancy; educational status, spousal relations, psycho-social support, family problems, presence of violence, and concerns about the baby. As a result of all these reasons, pregnancy hormones and neuroendocrine system are affected and cause nausea and vomiting. In addition, it is emphasized that unwanted pregnancy, perceived stress, acceptance of pregnancy are among the most important psychosocial factors that cause nausea and vomiting.

Pregnant women with nausea-vomiting may have feelings of isolation, loneliness, guilt, may consider terminating their pregnancy, and may experience anxiety about the effect of nausea-vomiting on their baby. Pregnant women experience anxiety for reasons such as not being able to concentrate on their baby, worrying about the future, adapting to pregnancy and thinking only about their own health, and the need for intervention for these parameters is increasing.

In psychoanalytic thought, nausea-vomiting during pregnancy is defined as a defense mechanism developed against unidentified discontent and the way the person expresses this situation. In order to change this discontent and the way of self-expression of the person, besides many psychotherapy methods, the emotional liberation technique, which is quick and easy to apply, and aims to reach the result in a short way by working on emotion-based, can have positive effects. Emotional liberation; It is an energy psychology technique that aims to free from negative emotions, clearing negative emotions, experiences, traumas and fears from the past and regulating the energy flow.

Energy psychology, which has thousands of years of history in eastern cultures and has been used in the treatment of psychological problems in the West for the last 40 years, is not that human consists of independent parts; It is a new method based on the holistic approach, which is believed to have the knowledge of the whole of each part. According to energy psychology, it is in harmony with human physiology, mental processes, emotions and behaviors. Along with these processes, human is considered as a whole, including the environment and culture. It hypothesizes that psychological disorders and other health conditions are associated with disturbances in the body's electrical energies and these energy fields, as well as congestion or disruption.

For this reason, emotional liberation technique, which is a non-pharmacological method, can be a practical method for psychological-based nausea-vomiting and anxiety by accepting the physiology, psychology, emotions and social environment of the pregnant as a whole.

ELIGIBILITY:
Inclusion Criteria:

* Not having a verbal communication problem,
* 6-12th of pregnancy be in the week
* Not having a psychiatric disorder
* Having a single, viable fetus
* Absence of a fetal congenital malformation
* Not having any disease other than pregnancy that will cause nausea and vomiting

Exclusion Criteria:

* Diagnosing a risky pregnancy during the research process,
* Asking to leave the research.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Subjective Units of Experience- (SUE) | Each participant will be evaluated for 1 week.
  The negative 10 feel the greatest pain, disappointment, fear, stress, sadness, or discomfort imaginable.
  When it reaches Positive 10, the client feels very different and wonderful. The meanings of the ratings in this range change gradually. The scale has no cutoff score. It is interpreted according to the mean of the scores and its relevance to other variables.

SECONDARY OUTCOMES:
Descriptive Data | It will be obtained in 1 month at the beginning of the research.
  Pregnant information form prepared by the researcher in line with the literature, socio-demographic (pregnant woman's age, education and employment status, income status, family type and place of residence), obstetric (current gestational week and pregnancy history), psycho-social and medical history (desire for pregnancy) status, whether there is a chronic disease) consists of questions.
Pregnancy Unique Quantification of Emesis and Nausea- (PUQE) | The time frame; pregnant women between 6 and 16 weeks included in the study will be evaluated for 4 weeks. It will take an average of 1 month to obtain the data. Measured PUQE scale data will be reported within 6 weeks at the end of the study.
  The PUQE test questions the number of nausea attacks, the number of vomiting, and the number of retching. A tight agreement was observed between the results obtained from the PUQE test and the Rhodes test (30). In the evaluation of the Puqe test, the total score was 3-6 as mild, 7-12 as moderate, and 13-15 as severe nausea and vomiting.
Pregnancy-Related Anxiety Questionnaire-2 (PRAQ-2) | The time frame; pregnant women between 6 and 16 weeks included in the study will be evaluated for 4 weeks. It will take an average of 1 month to obtain the data. Measured PRAQ-R2 scale data will be reported within 6 weeks at the end of the study.
  PRAQ-2 was developed by Van den Bergh in 1990 to measure the anxiety levels of women about their pregnancy periods and was revised by Huizink et al. It is a 5-point Likert-type scale, which was revised in 2016 to be applied to all pregnant women regardless of parity. It was adapted into Turkish by Aksoy Derya et al. The minimum and maximum scores that can be obtained from the scale are 11 and 55 for primiparas and 10 and 50 for multiparas, respectively. A score is calculated for each subscale of the PRAQ-2. As the score obtained from PRAQ-2 increases, the level of anxiety about pregnancy also increases. All statements in the questionnaire are positive statements. The scale does not have a breakpoint. The Cronbach's alpha reliability coefficient for the values calculated at various weeks of pregnancy was found to be between 0.71 and 0.85 in multiparas and between 0.75 and 0.84 in primiparas.

CONTACTS AND LOCATIONS:
Overall Officials: Zeliha OZSAHİN, Study Director — https://www.inonu.edu.tr/akademik/zeliha.ozsahin
Locations (1):
- Inonu University Faculty of Health Sciences Pregnant Education Class, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will be obtained with Personal Information Form, Subjective Experience Units (SUE), Pregnancy Unique Quantification of Emesis (PUQE) and Pregnancy-Related Anxiety Questionnaire - R2 (PRAQ-R2).

REFERENCES:
- [Derived] Guven Santur S, Ozsahin Z. The Effects of Emotional Freedom Techniques Implemented During Early Pregnancy on Nausea-Vomiting Severity and Anxiety: A Randomized Controlled Trial. J Integr Complement Med. 2024 Sep;30(9):858-868. doi: 10.1089/jicm.2023.0586. Epub 2024 Mar 27. PMID 38531058